CLINICAL TRIAL: NCT02490345
Title: Effect of Gabapentin on Postoperative Pain Control After a Cesarean Section
Brief Title: Gabapentin as Adjunctive Treatment for Postoperative Pain Control
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, David Haas, David Haas, MD, MS, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1507497375
Record Dates: First submitted 2015-07-01; First posted 2015-07-03 (Estimated); Last update posted 2017-08-23 (Actual); Status verified 2017-08

CONDITIONS: Drug Usage
Keywords: gabapentin
MeSH Terms: interventions — Gabapentin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gabapentin Administration (Active Comparator): gabapentin 600mg orally every 8 hours x 48 hours
  Interventions: Drug: gabapentin
- Placebo (Placebo Comparator): Placebo , 1 tablet, orally every 8 hours x 48 hours
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: gabapentin — gabapentin usage as adjunctive treatment for pain control
  Arms: Gabapentin Administration
Drug: Placebo — Identical placebo
  Arms: Placebo

SUMMARY:
The specific aims of this research study are to use 600 mg gabapentin as an adjunctive treatment for acute postoperative pain control in order to reduce postoperative opiate consumption and improve postoperative pain control.

DETAILED DESCRIPTION:
After consent has been obtained for the study and the cesarean has been completed, when the participant is in the recovery room, she will take the first pill of the study drug. This will occur approximately 30-60 minutes after the cesarean is completed. The time of first dose will be noted on the data capture form. The following will then occur:

* Participants will take study capsules (either 600 mg gabapentin or placebo) every 8 hours for the first 48 hours after beginning the study. The nurse on the unit will be sent the study drug in a blinded capsule by the Investigational Pharmacy.
* Participants will be asked about postoperative pain on a Visual Analog Scale by the care nurses or study personnel before each dose of study drug, before receiving any opioid medication, 2-4 hours after study drugs are consumed, at 24, 36 and 48 hours post surgery, and any other times during routine postoperative clinical care would warrant. Women record pain postoperatively on a similar scale as part of routine clinical care. Prescription pain medication will be given per clinical routine care. Study personnel will note how many pills were sent home.
* One week (6-9 days) after the cesarean delivery, participants will be contacted by phone or other preferred method and asked about pain score, somnolence scores, dizziness, nausea, depression, any problems they are experiencing, and asked how many pain pills are left in their prescriptions given when they went home. These data will be recorded.

An Edinburgh Depression Scale will also be administered upon consent, at 48 hours, and again at one week after delivery. If the scores meet the specified criteria, the provider will by notified or if the subject has already been discharged from the hospital, she will be given contact information for follow up care.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women at least 18 years of age
* Singleton gestation
* Gestational age equal to or greater than 30 weeks
* Women undergoing a non-emergent (often scheduled) repeat cesarean delivery
* Spinal anesthesia utilized during cesarean

Exclusion Criteria:

* History of opiate abuse
* Women on opiates during pregnancy
* Women requiring treatment with magnesium sulfate postpartum
* Preexisting Fibromyalgia, chronic pain syndrome, or rheumatologic disorder
* General anesthesia required for cesarean
* Plans to breastfeed
* History of major depression or postpartum depression requiring medication
* Planned classical cesarean section

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2015-10; Primary Completion 2017-06-29 (Actual); Study Completion 2017-06-29 (Actual)

PRIMARY OUTCOMES:
Amount of opioid equivalents consumed | 48 hours after cesarean delivery

SECONDARY OUTCOMES:
Amount of opioid equivalents consumed | one week after cesarean delivery
VAS pain scores | one week after cesarean delivery
Adverse events (somnolence, dizziness, nausea, depression, suicidal ideation, or notable peripheral edema) or drug reactions | one week after cesarean delivery

CONTACTS AND LOCATIONS:
Overall Officials: David Haas, MD, MS, Principal Investigator — Indiana School of Medicine
Locations (2):
- United States (2):
  - Eskenazi Health, Indianapolis, Indiana
  - Eskenazi Hospital, Indianapolis, Indiana

IPD SHARING:
Plan to Share IPD: Undecided